CLINICAL TRIAL: NCT05610072
Title: Glutamatergic Mechanisms in Opioid and Cocaine Co-Use
Brief Title: Behavioral Effects of Drugs (Inpatient): 43 (Opioids, Cocaine, n-Acetylcysteine)
Acronym: BED IN 43
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 80485; R33DA049130 (NIH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cocaine Use Disorder; Opioid Use Disorder; Stimulant Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Acetylcysteine; Hydromorphone

STUDY DESIGN:
Intervention Model Description: This study will use a double-blind, placebo-controlled design with all subjects receiving all hydromorphone (i.e., hydromorphone dose is a within subject factors). Half of the subjects will receive placebo and half of the subjects will receive 2.4mg/day NAC.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- n-Acetylcysteine (Experimental): Subjects will receive 0.6 g oral n-acetylcysteine 4 times per day.
  Interventions: Drug: n-acetylcysteine; Drug: Hydromorphone; Drug: Placebo hydromorphone
- Placebo (Placebo Comparator): Subjects will receive oral placebo 4 times per day.
  Interventions: Drug: Hydromorphone; Drug: Placebo n-acetylcystine; Drug: Placebo hydromorphone

INTERVENTIONS:
Drug: n-acetylcysteine — Subjects will be randomized to receive 2.4 oral n-acetylcysteine daily.
  Arms: n-Acetylcysteine
Drug: Hydromorphone — Subjects will receive up to 192 mg oral hydromorphone daily.
Drug: Placebo n-acetylcystine — Subjects will be randomized to receive placebo n-acetylcysteine daily.
  Arms: Placebo
Drug: Placebo hydromorphone — Prior to some experimental sessions, subjects will receive placebo hydromorphone

SUMMARY:
The overarching hypotheses of this protocol are that (1) persistent brain glutamate changes induced by chronic opioid use will exacerbate use of cocaine during opioid physical dependence and withdrawal and (2) n-acetylcysteine (NAC) will ameliorate glutamatergic dysregulation, and thus will reduce both opioid and cocaine demand. These hypotheses will be tested with two specific aims.

Specific Aim 1. Determine the reinforcing effects of cocaine in individuals with comorbid opioid and cocaine use disorder with physiological dependence on opioids during NAC maintenance. All subjects will be maintained on oral hydromorphone. They will also be randomly assigned to receive placebo or oral NAC (2.4 g/day), stratified by sex. After dose stabilization, experimental sessions will be conducted in which subjects complete hypothetical cocaine purchase tasks during opioid maintenance and opioid withdrawal. The hypotheses are: 1) cocaine purchasing will be greater during opioid withdrawal and 2) NAC maintenance will attenuate cocaine purchasing across opioid maintenance and withdrawal periods.

Specific Aim 2. Evaluate glutamate functionality during periods of opioid maintenance and withdrawal in individuals with comorbid opioid and cocaine use disorder and physiological dependence on opioids during NAC maintenance. Subjects will undergo magnetic resonance spectroscopy to evaluate brain glutamate changes as a function of opioid maintenance/withdrawal state and NAC maintenance. The hypotheses are: 1) glutamate levels will be elevated during opioid withdrawal and 2) NAC maintenance will ameliorate elevated glutamate levels.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 55 years,
2. Report recent use of opioids and cocaine and must not be seeking treatment for their drug use,
3. Be physically dependent on short-acting opioids,
4. Meet Diagnostic and Statistical Manual (DSM)-5 diagnostic criteria for current opioid use disorder (OUD) and current or past cocaine use disorder (CUD) and have either a urine sample positive for recent opioid use during each visit or if opioid negative, displaying frank withdrawal during screening
5. Other than the diagnosis for opioid and cocaine use disorder at the time of the screening, subjects must be healthy,
6. Laboratory chemistries (e.g., blood chemistry screen, complete blood count, urinalysis) and electrocardiogram (ECG) results must be normal or within normal range and any abnormal results must be considered as not clinically significant by the study physicians,
7. No contraindications to magnetic resonance imagining (MRI; e.g., metallic objects in their body, BMI > or = 40, claustrophobia) will be considered ineligible,
8. Female subjects must be using an effective form of birth control (e.g., birth control pills, surgical sterilization, intrauterine device, barrier method, condoms with spermicide, cervical cap with a spermicide or abstinence) to participate and must not be pregnant,
9. All study subjects will be judged by the medical staff to be psychiatrically and physically healthy.

Exclusion Criteria:

1. Any potential subject with a history of serious physical disease, current physical disease (e.g., impaired cardiovascular functioning, histories of seizure, head trauma, diabetes, asthma, or central nervous system [CNS] tumors) or current or past histories of serious psychiatric disorder (e.g., schizophrenia) that would limit compliance in the study, other than substance use disorder, will be excluded from research participation,
2. Potential subjects that meet diagnostic criteria for moderate - severe substance use disorder for substances other than opioids, stimulants, cannabis, or nicotine at the time of the interview will not be eligible for study participation,
3. Subjects who report a positive first-degree family history of schizophrenia, serious cardiovascular disease, or seizure disorders will also be excluded from research participation.
4. Subjects with contraindications to hydromorphone or n-acetylcysteine will not be eligible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypothetical opioid purchasing | After at least seven days of maintenance on n-acetylcysteine or placebo
  Amount of opioids purchased on a hypothetical purchase task
Hypothetical cocaine purchasing | After at least seven days of maintenance on n-acetylcysteine or placebo
  Amount of cocaine purchased on a hypothetical purchase task
Glutamate function | After at least seven days of maintenance on n-acetylcysteine or placebo
  Magnetic resonance spectroscopy of brain glutamate levels
Gamma Aminobutyric Acid (GABA) function | After at least seven days of maintenance on n-acetylcysteine or placebo
  Magnetic resonance spectroscopy of brain GABA levels

SECONDARY OUTCOMES:
Craving | After at least seven days of maintenance on n-acetylcysteine or placebo
  Scores on a locally developed craving scale from 1-10, with higher scores indicating more craving
Subjective opioid withdrawal | After at least seven days of maintenance on n-acetylcysteine or placebo
  Self-reported scores on the Subjective Opioid Withdrawal Scale with scores from 0-64, with higher scores indicating more withdrawal
Clinical opioid withdrawal | After at least seven days of maintenance on n-acetylcysteine or placebo
  Self-reported scores on the Clinical Opioid Withdrawal Scale with scores from 0-48, with higher scores indicating more withdrawal

OTHER OUTCOMES:
Side effects | Daily during approximately 10 day inpatient admission
  Scores on the Udvalg Fur Kliniske Undersolgelser (UKU) side effects scale with scores from 0-3, with higher scores indicating greater side effects
Pupil diameter | Daily during approximately 10 day inpatient admission
  Measurement of pupil diameter using an automated scanner
Heart rate | Daily during approximately 10 day inpatient admission
  Measurement of heart rate using an automated monitor
Respiration rate | Daily during approximately 10 day inpatient admission
  Measurement of respiration rate using an automated monitor
Oxygen saturation | Daily during approximately 10 day inpatient admission
  Measurement of oxygen saturation using an automated monitor
Diastolic blood pressure | Daily during approximately 10 day inpatient admission
  Measurement of diastolic blood pressure using an automated monitor
Systolic blood pressure | Daily during approximately 10 day inpatient admission
  Measurement of systolic blood pressure using an automated monitor

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky
  - University of Kentucky Department of Behavioral Science, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No